CLINICAL TRIAL: NCT04763109
Title: Identification of Pre-Malignant Lesions In Pediatric Patients With Neurofibromatosis Type 1 Using Novel Magnetic Resonance Imaging Techniques Paired With Artificial Intelligence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Baca (Other)
Responsible Party: Sponsor-Investigator, Nicole Baca, Assistant Professor of Department of Pediatrics, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IIT2020-23-BACA-MRINF1
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Neurofibromatosis Type 1
Keywords: Pediatric; Neurofibromatosis Type 1; magnetic resonance imaging
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Whole-Body Magnetic Resonance Imaging (Experimental)
  Interventions: Other: Whole-body Magnetic Resonance Imaging

INTERVENTIONS:
Other: Whole-body Magnetic Resonance Imaging — Whole-body Magnetic Resonance Imaging at baseline, 1 month, and 12 months

SUMMARY:
This is a single arm pilot trial of a novel whole-body Magnetic Resonance Imaging paired with artificial intelligence intervention, to evaluate feasibility defined as scan-rescan reliability, and to estimate the positive predictive value of changes in Magnetic Resonance Imaging scans from baseline to 12-month visit using an Artificial Intelligence algorithm, among 15 pediatric patients with neurofibromatosis type 1 at Cedars-Sinai Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 5 and <18 years at the start of study. If subject will turn 18 during the study, they will be allowed to enroll.
* Clinically or molecularly confirmed diagnosis of NF-1. Subjects with mosaic/segmental NF-1 also qualify for the study.

Exclusion Criteria:

* Requiring sedation for imaging.
* Implants and/or Devices: Mechanical, magnetic or electrical activated implants; Ferromagnetic implants and foreign bodies
* Claustrophobia, problems being in enclosed spaces, or inability to lie facing upwards.
* Allergy to animal dander or animal-instigated asthma.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
For scan re-scan reliability, utilize T2 imaging to evaluate the agreement between the baseline scan and the 1 Month scan, which is performed within 4 weeks of the baseline scan. | From Baseline to within 4 weeks of baseline
  T2 is a type of high-resolution multiparametric tissue mapping that measures quantitative metrics of the physical properties of tissue and allows comparison in longitudinal follow-up

SECONDARY OUTCOMES:
For change over time, the initial scan imaging using T1 and apparent diffusion coefficient (ACD) imaging, the baseline scan will be compared to the third scan, which is performed 12 months (+/- 3 months) after the baseline scan. | From Baseline to 12 months
  T1 and ACD is a type of high-resolution multiparametric tissue mapping that measures quantitative metrics of the physical properties of tissue and allows comparison in longitudinal follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Baca, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States